CLINICAL TRIAL: NCT02861105
Title: The Effect of LMWH on ICSI Outcome in Patients With Unexplained Infertility and Negative Immunological Markers; a Randomized Controlled Trial
Brief Title: The Effect of LMWH on ICSI in Patients With Unexplained Infertility and Negative Immunological Markers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mostafa Fouad Gomaa, Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASU-OG-333
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Unexplained Infertility
MeSH Terms: interventions — Heparin, Low-Molecular-Weight; Enoxaparin; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMWH supplementation (Active Comparator): 40 mg of enoxaparin injected subcutaneously every 24 hours starting the day of ovum pick-up to the documentation of fetal life by ultrasound at 7 weeks of gestation
  Interventions: Drug: LMWH
- 0.9% saline solution (Placebo Comparator): 0.9% saline injected subcutaneously every 24 hours starting the day of ovum pick-up to the documentation of fetal life by ultrasound at 7 weeks of gestation
  Interventions: Other: 0.9% saline solution

INTERVENTIONS:
Drug: LMWH — LMWH will be given on daily basis subcutaneously every 24 hours starting one day after ovum pick up till documentation of fetal life by ultrasound at 7 weeks.
  Other Names: Clexane; Enoxaparin
  Arms: LMWH supplementation
Other: 0.9% saline solution — 0.9% saline solution will be given subcutaneously every 24 hours starting one day after ovum pick up till documentation of fetal life by ultrasound at 7 weeks.
  Other Names: 0.9% sodium chloride solution
  Arms: 0.9% saline solution

SUMMARY:
The purpose of this study is to assess the efficacy of LMWH treatment in women with unexplained infertility and negative immunological markers undergoing ICSI.

DETAILED DESCRIPTION:
Inclusion criteria:

1. patients undergoing 1st trial ICSI
2. unexplained infertility
3. negative immunological markers including ACL abs, LAC, ANA, ATA, AnitdsDNA

Exclusion criteria:

1. previous IVF/ICSI
2. Any cause of infertility
3. Suspected and/or unexpected poor response during ovulation induction
4. positive immunological markers
5. Age > 40 years.

All participants will undergo IVF/ICSI cycle using the Long luteal phase protocol. the dose of gonadotropins will be calculated according to patient age and BMI. All patients will have 2-3 embryos transferred at D5 according to their age. the primary outcome will be LBR. secondary outcomes will include biochemical pregnancy rate and clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* age less than 38 years
* at least 12 months of infertility
* women with unexplained infertility

Exclusion Criteria:

* age more than or equals 38 years
* serum AMH level less than or equals 1 ng/ml
* patients of anticoagulant therapy
* immune-compromised patients
* patients with contraindications to low molecular weight heparin
* positive immunological markers
* patients with other than unexplained infertility
* male factor infertility
* refusal of participation
* patients with unexpected poor or over response during induction of ovulation

Max Age: 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 716 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Live birth Rate | at delivery

SECONDARY OUTCOMES:
Clinical Pregnancy Rate | at 7 weeks of gestation
Biochemical Pregnancy Rate | 14 days after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa F Gomaa, MD, Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: No